CLINICAL TRIAL: NCT00545311
Title: A Multi-Center, Randomized, Double-Blind, Parallel-Group Study to Investigate the Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of Multiple Inhaled NVA237 Doses at Four Dose Levels in COPD Patients
Brief Title: Safety and Tolerability of Multiple Inhaled NVA237 Doses in Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CNVA237A2103
Record Dates: First submitted 2007-10-15; First posted 2007-10-17 (Estimated); Last update posted 2008-01-08 (Estimated); Status verified 2007-12

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: multiple inhaled, NVA237, COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Glycopyrrolate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental): NVA237
  Interventions: Drug: NVA237
- 2 (Experimental): NVA237
  Interventions: Drug: NVA237
- 3 (Experimental): NVA237
  Interventions: Drug: NVA237
- 4 (Experimental): NVA237
  Interventions: Drug: NVA237
- 5 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NVA237
  Arms: 1
Drug: NVA237
  Arms: 2
Drug: NVA237
  Arms: 3
Drug: NVA237
  Arms: 4
Drug: Placebo
  Arms: 5

SUMMARY:
This study will evaluate the pharmacokinetics, pharmacodynamics and safety of multiple doses of the NVA237 in mild and moderate COPD patients .

ELIGIBILITY:
Inclusion Criteria:

* Male and/or female patients aged from 40-75 years of age with mild to moderate COPD.
* Diagnosis of mild/moderate COPD, according to the GOLD guidelines.
* Bronchodilatory response to ipratropium at screening
* Current or ex-smokers with a smoking history of >10 pack-years. Ten pack-years is defined as 20 cigarettes a day for 10 years, or 10 cigarettes a day for 20 years etc.
* Female patients must have been surgically sterilized at least 6 months prior to screening or: Postmenopausal women must have no regular menstrual bleeding for at least 1 year prior to inclusion.
* Lab and post-bronchodilator values within a certain range.
* Body mass index (BMI) must be within the range of 18 to 32 kg/m2.

Exclusion Criteria:

* Any significant medical condition that in the opinion of the Investigator may compromise patient safety, patient compliance, interfere with evaluations, or preclude completion of the trial.
* Any medical condition that may make spirometry unsafe
* History of glaucoma, symptomatic prostatism or urinary retention.
* Participation in any clinical investigation within 4 weeks prior to dosing or longer if required by local regulations and for any other limitation of participation based on local regulations. Previous participation in a study with either the investigational or comparator drugs does not exclude a patient from participation in this study.
* Donation or loss of 400 ml or more of blood within 8 weeks prior to first dosing, or longer if required by local regulation.
* Significant illness (other than respiratory illness) within the two weeks prior to dosing.
* Clinically significant ECG abnormalities indicative of an unstable underlying cardiac problem, e.g. recent myocardial infarction, 2nd/3rd degree heart block, or a family history grandparents, parents and siblings of a prolonged QT-interval syndrome.
* History of clinically significant drug allergy or history of atopic allergy (asthma, urticaria, eczematous dermatitis). A known hypersensitivity to the study drug or drugs similar to the study drug.
* History of immunocompromise, including a positive HIV (ELISA and Western blot) test result.
* A positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result.
* History of drug or alcohol abuse within the 12 months prior to dosing or evidence of such abuse as indicated by the laboratory assays conducted during the screening or baseline evaluations.
* Patients who are unable to demonstrate appropriate use of the Concept 1 device at screening

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-07; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) of NVA237 following single and repeated once-daily inhaled NVA237 doses

SECONDARY OUTCOMES:
-Pharmacodynamics (PD) and PK/PD relationships of NVA237 following single and repeated once-daily inhaled NVA237 doses -Safety and tolerability of NVA237 following single and repeated once-daily inhaled NVA237 doses

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Investigator site
Locations (4):
- Novartis Investigative site, Copenhagen, Denmark
- Germany (3):
  - Novartis investigative site, Berlin
  - Novartis investigative site, Mönchengladbach
  - Novartis Investigative Site, Munich